CLINICAL TRIAL: NCT03155152
Title: Decremental Exercise Protocol as a Training Stimulus: More or Less Efficient Than Traditional High-intensity Interval Training?
Brief Title: Decremental Exercise: a New Training Approach?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DECT_HIIT_2017
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-02

CONDITIONS: Exercise Performance of Fit Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DECT Group (Experimental): The DECT session consists of four bouts of 4 min high-intensity "decremental" exercise with 3 min of active recovery between bouts. Load is progressively decreased throughout each exercise bout. The training period will last for a total of 4 weeks, with three weekly sessions of supervised training
  Interventions: Other: DECT
- HIIT Group (Active Comparator): The HIIT session consists of four bouts of 4 min high-intensity "decremental" exercise with 3 min of active recovery between bouts. Load is kept constant throughout each exercise bout. The training period will last for a total of 4 weeks, with three weekly sessions of supervised training
  Interventions: Other: HIIT

INTERVENTIONS:
Other: DECT — The DECT program consists of a 4-week training intervention with three weekly sessions of high-intensity interval training, in which during each exercise bout the workload is imposed in a decremental fashion.
  Arms: DECT Group
Other: HIIT — The HIIT program consists of a 4-week training intervention with three weekly sessions of high-intensity interval training, in which during each exercise bout the workload is kept constant.
  Arms: HIIT Group

SUMMARY:
Different types of high-intensity interval training (HIIT) sessions are used by athletes in order to improve their physical performance, but innovative approaches to training are lacking. Therefore, in Part A of this study the physiological response to a standard HIIT and a new decremental exercise training (DECT) will be compared in runners and cyclists. Next, in Part B the training effects of a 4-week block of the HIIT and DECT will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* Healthy, i.e. normal physical and mental status (not taking any medication on a regular basis for more than a month, except contraceptive medication)
* Normal Body-Mass-Index (BMI): 18.5-24.9 kg·m-2
* Well-trained athletes: V̇O2max > 55.1 ml·min-1·kg-1 for men and > 50.1 ml·min-1·kg-1 for women
* Normal lung function
* Non-smoking
* Willing to adhere to the general study rules

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the same part (A or B) of the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Acute or chronic illness
* Intake of medications affecting performance or the respiratory, cardiovascular or neuromuscular system
* Insufficient training history (<3 yrs of participation in competitive cycling/running) or training volume (<40 km running/week or 150 km cycling/week) in the previous 6 months
* Recent (<3 months) history of orthopaedic injury or participation in structured high-intensity training blocks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Change in exercise performance | measured before and after the 4-week training block, during a time-trial (40 km cycling or 10 km running)
  Time taken to cover a fixed distance, in minutes

SECONDARY OUTCOMES:
Change in maximal oxygen uptake | Measured during a maximal incremental exercise test before and after the 4-week training block
  Measured in ml/kg/min
Average oxygen uptake | The two training session are performed within one week
  Average oxygen uptake measured during the four 4-min bouts of high-intensity exercise of a session of HIIT and DECT

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Spengler, Prof., Principal Investigator — ETH Zurich
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No